CLINICAL TRIAL: NCT03728478
Title: Comparison of STep-up and Step-down Therapeutic Strategies in Childhood ARthritiS
Brief Title: STep-up and Step-down Therapeutic Strategies in Childhood ARthritiS
Acronym: STARS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government); Compagnia di San Paolo (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Alessandro Consolaro, Principal Investigator, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-001931-27
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Oligoarthritis, Juvenile; Polyarthritis, Juvenile, Rheumatoid Factor Negative
Keywords: juvenile idiopathic arthritis; treatment; treat to target
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Intervention Model Description: This is a a 12-month open label, randomised, actively controlled, multi-centre, prospective, superiority trial of two different treatment strategies (Step-down versus Step-up).
  After signature of informed consent/assent patients will be randomized into two therapeutic arms: "Step-up" or "Step-down". Patients in the Step-up arm will be treated according to a conventional strategy based on treatment escalation and driven by the treat-to-target strategy. Patients in the Step-Down arm will be treated with an early, combined, aggressive therapy for 6 months.
  After the conclusion of the 12-month observation period of the trial, patients will be followed for up to 5 years for the evaluation of disease course, medication requirements, adverse events, and long-term disease-related morbidity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm 1: Step-up (No Intervention): JIA patients managed with a Treat-To-Target strategy (T2T)
- Treatment arm 2: Step-down (Experimental): JIA patients treated with an early combined therapy
  Interventions: Drug: Etanercept; Drug: Methotrexate; Drug: Intra-articular corticosteroid injections

INTERVENTIONS:
Drug: Etanercept — Patients will receive etanercept subcutaneously at a dose of 0.8 mg/kg weekly (up to a maximum dose of 50 mg weekly).
  Other Names: ETN
  Arms: Treatment arm 2: Step-down
Drug: Methotrexate — Methotrexate will be administered subcutaneously, in a single weekly dose of 15 mg/m2 (max 20 mg).
  Other Names: MTX
  Arms: Treatment arm 2: Step-down
Drug: Intra-articular corticosteroid injections — Triamcinolone hexacetonide and methylprednisolone acetate doses depend on the affected joint.
  Other Names: IACI
  Arms: Treatment arm 2: Step-down

SUMMARY:
This study aims to compare the effectiveness of a conventional therapeutic regimen, based on treatment escalation (step-up strategy) and driven by the treat-to-target approach, with that of an early aggressive intervention based on the initial start of a combination of conventional and biological DMARDs (step-down strategy).

DETAILED DESCRIPTION:
Although their approach is different, both interventions are aimed to obtain a quick and robust disease control and to maintain it over time. Compelling evidence exists that in children with chronic arthritis early intensive therapy may take advantage of the so-called "window of opportunity", in which the biology of the disease can be altered to improve long-term disease outcomes, including prevention of cumulative joint damage. Recent experiences in children with systemic JIA have shown that early anti-IL-1 therapy may lead to rapid achievement of inactive disease and allow early treatment discontinuation without disease relapses in many patients. The benefits of early treatment with biologic agents in other JIA categories are less clear, but convincing evidence has been recently reported for polyarthritis.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all the following criteria in order to be enrolled in the trial:

I. Newly-diagnosed and synthetic or biologic DMARD-naïve children (only treatment with 1 NSAID is allowed and no corticosteroid joint injections prior to randomization ) with a JIA classified according to the following ILAR categories:

i. Oligoarthritis ii. Rheumatoid factor negative polyarthritis

II. Active arthritis

III. Onset of JIA symptoms no more than 6 months before randomization

IV. Age 2 to 17 years at enrolment.

V. Female of child-bearing potential must have a negative pregnancy test at the beginning of the trial. If sexually active, they must agree to use highly effective contraceptive measures, throughout study participation, and must have no intention of conceiving during the course of the study. Post-pubertal males must have no plans to father a child during the study and agree to use highly effective contraceptive measures if sexually active.

VI. Ability to comply with the entire study procedures, ability to communicate meaningfully with the investigational staff, competence to give written informed consent; to be applied to the parents and/or patients, as appropriate

VII. Duly executed, written, informed consent/assent obtained from the parents/patient.

Exclusion criteria

I. Classification in one of the following JIA categories: systemic arthritis, RF-positive polyarthritis, psoriatic arthritis, enthesitis-related arthritis, undifferentiated arthritis

II. Patients who need systemic treatment for uveitis

III. Tuberculosis related issues: patients are excluded from the study if they have:

1. Active TB or a history of incompletely treated TB
2. PPD or QuantiFERON-TB positive patients (with no active disease) unless it is documented by a specialist that the patient has been adequately treated for TB and can start treatment with a biologic agent, based on the medical judgment of the study investigator and / or an infectious disease specialist.
3. Suspected extrapulmonary TB infection
4. Patients at high risk of contracting TB, such as close contact with individual with active or latent TB

IV. Previous treatment with any synthetic or biologic DMARD

V. Any live attenuated vaccine within 4 weeks prior to the baseline visit, such as varicella-zoster, oral polio, measles, mumps or rubella vaccines and throughout the study. Killed or inactive vaccine may be permitted based on the investigator's judgment

VI. Prior or current history of malignancy or any other significant concomitant illness(es) as per the treating physician evaluation

VII. Any of the following laboratory abnormalities based on the most recent laboratory results:

1. White blood cell (WBC) count <3.50 x 103/mm3 (SI units: <3.50 x 109/L) and neutrophils < 1x109/L;
2. Hemoglobin < 8.5 g/dL (SI units: <85 g/L);
3. Platelet Count < 125,0000/mm3 or ≥1,000,000/mm3 (SI units: <125 x 109/L or ≥1,000 x 109/L
4. Aspartate aminotransaminase (AST) or alanine aminotransaminase (ALT) ≥ 2.0 x upper limit of normal (ULN).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical remission on or off medication at 12 months | 12 months
  The effectiveness of the two therapeutic strategies will be compared by assessing the frequency of clinical remission (CR) at 12 months. CR is defined as the persistence of the JADAS state of ID for at least 6 months.

SECONDARY OUTCOMES:
Inactive disease | 12 months
  The rate of patients who achieve the JADAS/JIA ACR state of ID at any single point in time throughout the study period will be compared between the 2 arms.
Time to inactive disease as per JADAS/JIA ACR criteria | 12 months
  Time to achieve the state of JADAS/JIA ACR ID will be calculated as the time difference (in days) between the date of randomization and the date of the visit at which the patient will be observed to be in ID.
Time to JADAS/JIA ACR clinical remission | 12 months
  Time to achieve the state of JADAS/JIA ACR ID will be calculated as the time difference (in days) between the date of randomization and the date of the visit at which the patient will be observed to be in clinical remission (i.e. persistent inactive disease for at least 6 months).
Time spent in JADAS/JIA ACR inactive disease | 12 months
  The cumulative time spent in the JADAS/JIA ACR state of ID will be calculated as the time difference (in days) between the date of the first visit at which the patient will be observed to be in ID and the date at which he/she will be observed to be no longer in ID that is when the disease will flare (see later for definitions), or database closure for analysis purposes. We will assume that if a patient is found to be in ID at 2 consecutive visits, the patient had ID on all days between these visits. If a patient will be found to have ID at a particular visit, but lost the ID status at the subsequent visit, the patient will be considered to have been in ID until the recurrence of active disease. Patients found to be in ID only at the time of database closure will contribute a single day of ID. The time in inactive disease per patient will be recorded and compared between the 2 arms.
Cumulative level of disease activity throughout the study period | 12 months
  The area under the curve (AUC) of the JADAS10 score assessed at every study visit and the AUC of the parent version of the JADAS (parJADAS) assessed monthly will be recorded and compared between the 2 arms.
Time spent on therapy | 12 months
  The cumulative time on therapy will be calculated as the time difference (in days) between the date of the visit at which the patient will start a systemic medication (synthetic or biologic DMARDs or steroids) until the date at which he/she will be observed to no longer be in treatment with a systemic medication, or completed the study. We assume that if a patient does not receive medications at 2 consecutive visits, the patient had not received medications all days between these visits. Patients initiating a systemic treatment at the final visit of the study will contribute a single day of time in therapy. The mean percentage of time spent on therapy per patient will be recorded and compared between the 2 arms.
Rate of flares | 12 months
  The rate of patients who develop flare, defined as the recurrence of active disease after attaining inactive disease at last visit according JADAS or JIA ACR definition, and the number of flares and the time to flare per patient will be recorded and compared. Notably, all patients prescribed intra-articular injections, synthetic or biologic DMARDs or systemic steroids will be considered as flare independently from JADAS or ACR criteria.
Rate of uveitis onset | 12 months
  The rate of patients who develop uveitis according to the Standardized Uveitis Nomenclature (SUN) will be recorded and compared between the 2 arms. The rate of patients requiring systemic medications for treatment of uveitis will be also recorded and compared between the 2 arms. However, these patients will be excluded from the study and followed for safety only.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Giannina Gaslini, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallace CA, Giannini EH, Spalding SJ, Hashkes PJ, O'Neil KM, Zeft AS, Szer IS, Ringold S, Brunner HI, Schanberg LE, Sundel RP, Milojevic D, Punaro MG, Chira P, Gottlieb BS, Higgins GC, Ilowite NT, Kimura Y, Hamilton S, Johnson A, Huang B, Lovell DJ; Childhood Arthritis and Rheumatology Research Alliance. Trial of early aggressive therapy in polyarticular juvenile idiopathic arthritis. Arthritis Rheum. 2012 Jun;64(6):2012-21. doi: 10.1002/art.34343. Epub 2011 Dec 19. PMID 22183975
- [Background] Ravelli A, Consolaro A, Horneff G, Laxer RM, Lovell DJ, Wulffraat NM, Akikusa JD, Al-Mayouf SM, Anton J, Avcin T, Berard RA, Beresford MW, Burgos-Vargas R, Cimaz R, De Benedetti F, Demirkaya E, Foell D, Itoh Y, Lahdenne P, Morgan EM, Quartier P, Ruperto N, Russo R, Saad-Magalhaes C, Sawhney S, Scott C, Shenoi S, Swart JF, Uziel Y, Vastert SJ, Smolen JS. Treating juvenile idiopathic arthritis to target: recommendations of an international task force. Ann Rheum Dis. 2018 Jun;77(6):819-828. doi: 10.1136/annrheumdis-2018-213030. Epub 2018 Apr 11. PMID 29643108
- [Derived] Tan J, Renton WD, Whittle SL, Takken T, Johnston RV, Tiller G, Munro J, Buchbinder R. Methotrexate for juvenile idiopathic arthritis. Cochrane Database Syst Rev. 2024 Feb 9;2(2):CD003129. doi: 10.1002/14651858.CD003129.pub2. PMID 38334147
- [Derived] Burrone M, Mazzoni M, Naddei R, Pistorio A, Spelta M, Scala S, Patrone E, Garrone M, Lombardi M, Villa L, Pascale G, Cavanna R, Ruperto N, Ravelli A, Consolaro A; Paediatric Rheumatology International Trials Organisation (PRINTO). Looking for the best strategy to treat children with new onset juvenile idiopathic arthritis: presentation of the "comparison of STep-up and step-down therapeutic strategies in childhood ARthritiS" (STARS) trial. Pediatr Rheumatol Online J. 2022 Sep 7;20(1):80. doi: 10.1186/s12969-022-00739-x. PMID 36071444